CLINICAL TRIAL: NCT01836484
Title: Diagnostic Accuracy of MRI, Diffusion-weighted MRI, FDG-PET/CT and Fluoro-ethyl-choline PET/CT in the Detection of Lymph Node Metastases in Surgically Staged Endometrial and Cervical Carcinoma
Brief Title: Diagnostic Accuracy of MRI, DWI MRI, FDG-PET/CT and FEC PET/CT in the Detection of Lymph Node Metastases in Surgically Staged Endometrial and Cervical Carcinoma
Acronym: MAPPING
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Birmingham Women's NHS Foundation Trust (Other Government); Case Western Reserve University (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Hammersmith Hospitals NHS Trust (Other); Memorial Sloan-Kettering Cancer Center, USA (Unknown); Queen Elizabeth Hospital, Gateshead, UK (Unknown); Royal Preston Hospital, Lancashire, UK (Unknown); Royal Marsden NHS Foundation Trust (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 007697
Record Dates: First submitted 2013-01-31; First posted 2013-04-22 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Surgically Staged Endometrial and Cervical Carcinoma; Cervical Cancer: Invasive Disease, FIGO Stage 1B1 or Higher; Endometrial Cancer; Stage 1A With Myometrial Invasion or Any Higher Stage and Grade 3; Stage 1A With Myometrial Invasion or Any Other Higher Stage and Serous Papillary or Clear Cell Sub-types; Stage II Disease or Above and Any Histology Grade
Keywords: Surgically staged endometrial carcinoma; Surgically staged cervical carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Lymphoma, Follicular; Disease | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Lymph node tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgically staged endometrial and cervical carcinoma
  Interventions: Diagnostic Test: Diffusion-weighted MRI; Diagnostic Test: Fluorodeoxyglucose-18-PET/CT; Diagnostic Test: Fluoro-ethyl-coline-PET/CT

INTERVENTIONS:
Diagnostic Test: Diffusion-weighted MRI
  Other Names: DW-MRI
Diagnostic Test: Fluorodeoxyglucose-18-PET/CT
  Other Names: FDG-PET/CT
Diagnostic Test: Fluoro-ethyl-coline-PET/CT
  Other Names: FEC-PET/CT

SUMMARY:
This is a prospective diagnostic performance study which compares three new imaging methods with the current standard imaging method for the diagnosis of metastatic lymph nodes.

DETAILED DESCRIPTION:
The aim is to demonstrate whether leading edge molecular imaging technologies (FDG-PET/CT, DW-MRI and Fluoro-ethyl-choline (FEC) PET/CT) can identify lymph node metastases with sufficient accuracy to allow non-invasive lymph node staging in patients with endometrial and cervical carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years or older; (no upper limit).
2. Patients with histologically confirmed cancer of the cervix or endometrium.

   1. In patient with cervix cancer, there must be confirmation of invasive disease; FIGO stage 1B1 or higher FIGO stage demonstrated clinically and/or on MRI. In patients with advanced disease being considered for chemoradiotherapy treatment, patients may be considered for entry if nodal lymphadenectomy is being used to inform radiotherapy planning;
   2. In patients with endometrial cancer, a) stage 1A with myometrial invasion or any higher stage and grade 3 b) stage 1A with myometrial invasion or any other higher stage and serous papillary or clear cell sub-types
   3. stage II disease or above and any histology grade The MDT decision may be based on the combination of tumour characteristics on histology, clinical and imaging findings.
3. No contra-indication to FDG-PET/CT, FEC-PET/CT or MRI.
4. Fit for surgical lymphadenectomy, as determined by the local MDT. The patient should also be considered fit for extended field radiotherapy in cases where lymphadenectomy is being undertaken to inform radiotherapy planning.

   The extent of lymph node dissection will be made by the local multidisciplinary team, based on the presence of risk factors for lymph node metastases, according to the protocol. Patients must be considered fit to undergo lymph node dissection.
5. Able and willing to give written informed consent and to comply with the study protocol procedures

Exclusion Criteria:

1. Known contra-indication to MRI or PET/CT scan.
2. Known allergy to FDG or FEC.
3. Not considered fit for lymphadenectomy (open or laparoscopic) or, where appropriate, radiotherapy, as determined by the local MDT.
4. If the patient is pregnant or breast-feeding.
5. Females of childbearing potential must be willing to use an effective method of contraception (hormonal or barrier method of birth control) from the time consent is signed until 6 weeks after the last PET/CT scan unless undergoing hysterectomy.

   Note: subjects are not considered of childbearing potential if they are surgically sterile (they have undergone bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal
6. Females of childbearing potential must have a negative pregnancy test within three weeks prior to being registered for the study.
7. Participation in another Clinical Trial of an Investigational Medicinal Product (CTIMP). If patient's have recently completed a CTIMP trial they must have had their last dose(s) of study drug prior to their first imaging procedure on the MAPPING study.
8. Participation in another clinical trial (CTIMP or non-CTIMP) where the protocol contains imaging procedures that would occur during the MAPPING study.
9. Medical or psychiatric illness, which makes the patient unsuitable or unable to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 women with histologically confirmed endometrial or cervical carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Detection rate (DR) vrs false positive rate (FPR) for each of the diagnostic modalities. | 36 months

SECONDARY OUTCOMES:
Detection rate (DR) vrs false positive rate (FPR) between each of the diagnostic modalities and within different histological sub-sets. | 36 months
Nodal Coverage planning: standard radiotherapy planning vrs DW-MRI | 36 months
Histopathological findings vrs functional imaging findings | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rockall, Professor, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (7):
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham University Hospitals, Birmingham NHS Foundation Trust, Birmingham
  - Birmingham City Hospital, Sandwell & West Birmingham Hospitals NHS Trust, Birmingham
  - St Bartholomew's Hospital, Barts Health NHS Trust, London
  - University College London Hospital, London
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Royal Preston Hospital, Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - The Royal Marsden, The Royal Marsden NHS Foundation Trust, Sutton